CLINICAL TRIAL: NCT00186277
Title: Phase II Study of Oxaliplatin and Taxotere in Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sandy Srinivas, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLDR0001; BLDR0001 (Other: Stanford University)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oxaliplatin — Calculated per patient
  Other Names: Eloxatin
Drug: Taxotere — Calculated per patient
  Other Names: Docetaxel

SUMMARY:
To combine oxaliplatin and taxotere in patients who have had prior cisplatin therapy in bladder cancer.

DETAILED DESCRIPTION:
To test the combination of oxaliplatin chemotherapy in combination with taxotere chemotherapy in patients with advanced bladder cancer who have failed one prior chemotherapy.

ELIGIBILITY:
* Patient Population Type: Advanced Muscle Invasive Bladder Cancer
* Prior Therapy: One prior therapy for advanced disease
* Disease: Measurable disease
* ECOG Performance: 0,1
* Indication: Histologically Proven Carcinoma of the bladder
* For female patient of childbearing potential, neither pregnant nor breastfeeding, and under active contraception
* Allergies: No known allergy to one of the study drugs
* Patient Status:
* No CNS metastases
* No peripheral neuropathy > grade1
* No other serious concomitant illness
* Fully recovered from any prior therapy
* Informed Consent: Patient and doctor have signed informed consent
* Lower Age Limit: Lower age limit >18
* Upper Age Limit: Upper Age Limit <70
* ANC: ANC >1500/mm3 or WBC > 3000/mm3
* Platelets: Platelets >100,000/mm3
* Creatinine: Creatinine <1.8mg/dL
* Bilirubin: Bilirubin <=2.0 x ULN
* SGPT: SGPT (ALT) <=1.5 x ULN (<4xULN if liver metastases present)
* RBC: Hemoglobin > 9.0g/dL
* Cardiovascular: No active congestive heart failure, no uncontrolled angina, no myocardial infarction within the past 6 months
* Patients with metastatic cancer of the urothelial tract (TCC, Adenocarcinoma)
* No prior exposure to Oxaliplatin
* No cytotoxics or radiation 4 weeks prior to enrolling on protocol
* PT/PTT normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Tolerability of the this combination in patients with recurrent metastatic bladder cancer. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States